CLINICAL TRIAL: NCT03259022
Title: Bronchial Infection in Patients With COPD and Frequent Exacerbations; Role of Innate Immunity and the Use of an Electronic Nose for Diagnosis.
Brief Title: Bronchial Infection in Patients With COPD and Frequent Exacerbations.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-BRO-2015-92
Record Dates: First submitted 2016-09-07; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Quantitative sputum culture, oral lavage, peripheral blood and exhaled air intake will be conducted.
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis:

1. Innate immunity is altered in certain patients with COPD and frequent exacerbations, a fact that makes them more susceptible to being infected by bacteria.
2. The electronic nose is able to detect patterns of specific VOCs for exacerbations of infectious origin.

DETAILED DESCRIPTION:
Bronchial infection has been described as the leading cause of COPD exacerbations. Different studies with invasive endoscopic techniques have demonstrated the presence of bacteria in the air in 40-70% of exacerbations of the disease. In addition, these patients have a higher concentration of cells and proinflammatory cytokines in the airway. This increased inflammation is associated with more frequent and more severe exacerbations, which worsen this vicious circle.

It is not known why some patients with COPD are more susceptible than others to bronchial, acute or chronic infection. Recent studies have suggested the importance of lung innate immunity, both humoral (proteins with antibiotic activity, inflammatory mediators) and cell (neutrophils, macrophages) as the key to the defense of the lung against infectious agents external factor. There may be a bidirectional relationship between immune response and bronchial infection in COPD exacerbations.

Te main objectives of our study are: 1. To study the expression of mucin, PAM and TLR in the airway of patients with COPD and frequent exacerbations (FE) and its relationship with the infection of the airway. 2. Determine the patterns of volatile organic compounds (VOCs) detected by electronic nose associated with bronchial infection in patients with COPD and FE.

Secondary objectives: 1. To study the relationship between the expression of mucin, PAM and TLR with pulmonary and systemic inflammation. 2. To study the relationship between the expression of mucin, PAM and TLR with bronchial bacterial load. 3. To study the expression of mucin, PAM and TLR at the time of COPD exacerbations and subsequent clinical phase stability. 4. Determine VOC patterns for specific pathogens (H. influenzae, S. pneumoniae, P. aeurginosa). 5. To study the time evolution of patterns of VOCs after a COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of COPD according to national and international guidelines.
2. Presence of ≥ 2 exacerbations requiring admission in the last 12 months.
3. Signature of informed consent.

Exclusion criteria:

1. Presence of other lung diseases
2. terminal concomitant disease

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients with frequent exacerbations.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Relationship between infection and airway innate immunity of patients with COPD and frequent exacerbations. | 6 months
  Mucine levels will be determined with ELISA kits
Association between volatile organic compounds (VOCs) detected by an electronic nose and bronchial infection in patients with COPD and frequent exacerbations. | 6 months
  The patterns of specific volatile organic compounds in echaled air will be determined with electronic nose device.

SECONDARY OUTCOMES:
Relationship between airway innate immunity and systemic inflammation. | 6 months
  Mucin levels will be determined with ELISA kits
Relationship between airway innate immunity and bronchial bacterial load. | 6 months
  Mucin levels will be determined with ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Sibila, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Miravitlles M, Soler-Cataluna JJ, Calle M, Molina J, Almagro P, Quintano JA, Riesco JA, Trigueros JA, Pinera P, Simon A, Rodriguez-Hermosa JL, Marco E, Lopez D, Coll R, Coll-Fernandez R, Lobo MA, Diez J, Soriano JB, Ancochea J. Spanish guideline for COPD (GesEPOC). Update 2014. Arch Bronconeumol. 2014 Jan;50 Suppl 1:1-16. doi: 10.1016/S0300-2896(14)70070-5. No abstract available. PMID 24507959
- [Background] Anzueto A, Sethi S, Martinez FJ. Exacerbations of chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2007 Oct 1;4(7):554-64. doi: 10.1513/pats.200701-003FM. PMID 17878469
- [Background] Seemungal TA, Donaldson GC, Bhowmik A, Jeffries DJ, Wedzicha JA. Time course and recovery of exacerbations in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2000 May;161(5):1608-13. doi: 10.1164/ajrccm.161.5.9908022. PMID 10806163
- [Background] Soler-Cataluna JJ, Martinez-Garcia MA, Roman Sanchez P, Salcedo E, Navarro M, Ochando R. Severe acute exacerbations and mortality in patients with chronic obstructive pulmonary disease. Thorax. 2005 Nov;60(11):925-31. doi: 10.1136/thx.2005.040527. Epub 2005 Jul 29. PMID 16055622
- [Background] Wedzicha JA, Seemungal TA. COPD exacerbations: defining their cause and prevention. Lancet. 2007 Sep 1;370(9589):786-96. doi: 10.1016/S0140-6736(07)61382-8. PMID 17765528
- [Background] Hurst JR, Vestbo J, Anzueto A, Locantore N, Mullerova H, Tal-Singer R, Miller B, Lomas DA, Agusti A, Macnee W, Calverley P, Rennard S, Wouters EF, Wedzicha JA; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Susceptibility to exacerbation in chronic obstructive pulmonary disease. N Engl J Med. 2010 Sep 16;363(12):1128-38. doi: 10.1056/NEJMoa0909883. PMID 20843247
- [Background] Soler N, Ewig S, Torres A, Filella X, Gonzalez J, Zaubet A. Airway inflammation and bronchial microbial patterns in patients with stable chronic obstructive pulmonary disease. Eur Respir J. 1999 Nov;14(5):1015-22. doi: 10.1183/09031936.99.14510159. PMID 10596683
- [Background] Sethi S, Murphy TF. Infection in the pathogenesis and course of chronic obstructive pulmonary disease. N Engl J Med. 2008 Nov 27;359(22):2355-65. doi: 10.1056/NEJMra0800353. No abstract available. PMID 19038881
- [Background] Mizgerd JP. Respiratory infection and the impact of pulmonary immunity on lung health and disease. Am J Respir Crit Care Med. 2012 Nov 1;186(9):824-9. doi: 10.1164/rccm.201206-1063PP. Epub 2012 Jul 12. PMID 22798317
- [Background] Roy MG, Livraghi-Butrico A, Fletcher AA, McElwee MM, Evans SE, Boerner RM, Alexander SN, Bellinghausen LK, Song AS, Petrova YM, Tuvim MJ, Adachi R, Romo I, Bordt AS, Bowden MG, Sisson JH, Woodruff PG, Thornton DJ, Rousseau K, De la Garza MM, Moghaddam SJ, Karmouty-Quintana H, Blackburn MR, Drouin SM, Davis CW, Terrell KA, Grubb BR, O'Neal WK, Flores SC, Cota-Gomez A, Lozupone CA, Donnelly JM, Watson AM, Hennessy CE, Keith RC, Yang IV, Barthel L, Henson PM, Janssen WJ, Schwartz DA, Boucher RC, Dickey BF, Evans CM. Muc5b is required for airway defence. Nature. 2014 Jan 16;505(7483):412-6. doi: 10.1038/nature12807. Epub 2013 Dec 8. PMID 24317696
- [Background] Thornton DJ, Rousseau K, McGuckin MA. Structure and function of the polymeric mucins in airways mucus. Annu Rev Physiol. 2008;70:459-86. doi: 10.1146/annurev.physiol.70.113006.100702. PMID 17850213
- [Background] Kirkham S, Kolsum U, Rousseau K, Singh D, Vestbo J, Thornton DJ. MUC5B is the major mucin in the gel phase of sputum in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Nov 15;178(10):1033-9. doi: 10.1164/rccm.200803-391OC. Epub 2008 Sep 5. PMID 18776153
- [Background] Fujisawa T, Chang MM, Velichko S, Thai P, Hung LY, Huang F, Phuong N, Chen Y, Wu R. NF-kappaB mediates IL-1beta- and IL-17A-induced MUC5B expression in airway epithelial cells. Am J Respir Cell Mol Biol. 2011 Aug;45(2):246-52. doi: 10.1165/rcmb.2009-0313OC. Epub 2010 Oct 8. PMID 20935193
- [Background] Yang D, Biragyn A, Hoover DM, Lubkowski J, Oppenheim JJ. Multiple roles of antimicrobial defensins, cathelicidins, and eosinophil-derived neurotoxin in host defense. Annu Rev Immunol. 2004;22:181-215. doi: 10.1146/annurev.immunol.22.012703.104603. PMID 15032578
- [Background] Harder J, Meyer-Hoffert U, Teran LM, Schwichtenberg L, Bartels J, Maune S, Schroder JM. Mucoid Pseudomonas aeruginosa, TNF-alpha, and IL-1beta, but not IL-6, induce human beta-defensin-2 in respiratory epithelia. Am J Respir Cell Mol Biol. 2000 Jun;22(6):714-21. doi: 10.1165/ajrcmb.22.6.4023. PMID 10837369
- [Background] Parameswaran GI, Sethi S, Murphy TF. Effects of bacterial infection on airway antimicrobial peptides and proteins in COPD. Chest. 2011 Sep;140(3):611-617. doi: 10.1378/chest.10-2760. Epub 2011 Feb 24. PMID 21349930
- [Background] Medzhitov R. Toll-like receptors and innate immunity. Nat Rev Immunol. 2001 Nov;1(2):135-45. doi: 10.1038/35100529. PMID 11905821
- [Background] Berenson CS, Wrona CT, Grove LJ, Maloney J, Garlipp MA, Wallace PK, Stewart CC, Sethi S. Impaired alveolar macrophage response to Haemophilus antigens in chronic obstructive lung disease. Am J Respir Crit Care Med. 2006 Jul 1;174(1):31-40. doi: 10.1164/rccm.200509-1461OC. Epub 2006 Mar 30. PMID 16574934
- [Background] Berenson CS, Kruzel RL, Eberhardt E, Dolnick R, Minderman H, Wallace PK, Sethi S. Impaired innate immune alveolar macrophage response and the predilection for COPD exacerbations. Thorax. 2014 Sep;69(9):811-8. doi: 10.1136/thoraxjnl-2013-203669. Epub 2014 Mar 31. PMID 24686454
- [Background] Vidal S, Bellido-Casado J, Granel C, Crespo A, Plaza V, Juarez C. Flow cytometry analysis of leukocytes in induced sputum from asthmatic patients. Immunobiology. 2012 Jul;217(7):692-7. doi: 10.1016/j.imbio.2011.11.008. Epub 2011 Dec 2. PMID 22204819
- [Background] Buszewski B, Kesy M, Ligor T, Amann A. Human exhaled air analytics: biomarkers of diseases. Biomed Chromatogr. 2007 Jun;21(6):553-66. doi: 10.1002/bmc.835. PMID 17431933
- [Background] Hanson CW 3rd, Thaler ER. Electronic nose prediction of a clinical pneumonia score: biosensors and microbes. Anesthesiology. 2005 Jan;102(1):63-8. doi: 10.1097/00000542-200501000-00013. PMID 15618788
- [Background] Fens N, Zwinderman AH, van der Schee MP, de Nijs SB, Dijkers E, Roldaan AC, Cheung D, Bel EH, Sterk PJ. Exhaled breath profiling enables discrimination of chronic obstructive pulmonary disease and asthma. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1076-82. doi: 10.1164/rccm.200906-0939OC. Epub 2009 Aug 27. PMID 19713445
- [Background] Sibila O, Garcia-Bellmunt L, Giner J, Merino JL, Suarez-Cuartin G, Torrego A, Solanes I, Castillo D, Valera JL, Cosio BG, Plaza V, Agusti A. Identification of airway bacterial colonization by an electronic nose in Chronic Obstructive Pulmonary Disease. Respir Med. 2014 Nov;108(11):1608-14. doi: 10.1016/j.rmed.2014.09.008. Epub 2014 Sep 19. PMID 25269711